CLINICAL TRIAL: NCT00208962
Title: Allogeneic Cell Therapy for Adults With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amelia A Langston, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000722
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Hematologic Diseases
Keywords: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Procedure: chemotherapy and blood stem cell transplantation

INTERVENTIONS:
Procedure: chemotherapy and blood stem cell transplantation — A combination of conventional dose chemotherapy, granulocyte-colony stimulating factor (G-CSF) mobilized HLA-identical related allogeneic PBSC transplant, and post transplant infusions of donor leukocytes.

SUMMARY:
This is a research study involving the treatment of leukemia or lymphoma (lymph gland cancer) in adults who have leukemia or lymphoma that is unlikely to be cured with regular anticancer drugs or radiation treatments.

DETAILED DESCRIPTION:
This is a research study involving the treatment of leukemia or lymphoma (lymph gland cancer) in adults who have leukemia or lymphoma that is unlikely to be cured with regular anticancer drugs or radiation treatments. Intensive treatment with high doses of chemotherapy followed by a bone marrow transplant (BMT) from an HLA-(tissue-type) matched related donor would provide the best chance for cure of this leukemia or lymphoma. However, the success of BMT from relatives is limited in patients who are older than 50 years and/or have organ dysfunction by substantial complications due to the high dose chemotherapy related toxicity, graft-versus- host disease (GVHD), and relapse. Patients eligible for this study have an HLA matched sibling, but a BMT from the sibling would carry a high risk for severe side effects due to the patient's age, and/or organ dysfunction.

Researchers are evaluating a new treatment for adult patients with leukemia and lymphoma which involves regular dose chemotherapy and blood stem cell transplantation from an HLA-matched relative, with injections of donor immune cells (a type of white blood cells) given if you later relapse. In this study, the safety and feasibility of this treatment strategy are being investigated.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible as a recipient for this study, patients must have chronic myelocytic leukemia (CML) in chronic phase and be older than 60 years of age, have advanced myelodysplastic syndrome (MDS) and be over 60 years of age, have chronic lymphocytic leukemia (CLL) and be over 50 years of age, or have low grade lymphoma and be over 50 years of age. HLA typing of the recipient's family will be used to identify potential donors. Please contact study nurse for additional eligibility criteria. Final eligibility will be determined by the health professionals conducting this clinical trial.

Exclusion Criteria:

* Patients with an active, invasive/systemic fungal infection and patients with serologic evidence of antibodies to HIV I/II will be excluded from participating as recipients in this study. Additional exclusion factors include: patients who are pregnant or lactating, those with active central nervous system (CNS) malignant disease, and patients whose life expectancy is limited by diseases other than the disease for which the transplant is being performed. Please contact study nurse for additional ineligibility criteria. Final eligibility will be determined by the health professionals conducting this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1998-09; Primary Completion 2007-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Determine if conventional dose chemotherapy followed by allogeneic peripheral blood stem cell (PBSC) transplant and short course immunosuppression provide stable, sustained mixed donor-host chimerism. | 100 days

SECONDARY OUTCOMES:
Determine degree of donor-derived hematopoiesis and disease status on day +21, +40, +90, +140, and 180; overall survival and disease free survival at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Langston, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States